CLINICAL TRIAL: NCT05185492
Title: Multi-center Collaborative to Enhance Quality and Outcomes in the Management of Cardiogenic Shock
Acronym: VANQUISH SHOCK
Status: Recruiting | Type: Observational
Sponsor: STAVROS G DRAKOS (Other)
Responsible Party: Sponsor-Investigator, STAVROS G DRAKOS, Professor, Internal Medicine, University of Utah
Organization: University of Utah (Other)
Other Study IDs: IRB_00148867
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cardiogenic Shock; Acute Myocardial Infarction
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiogenic shock cohort: Primary diagnosis of Cardiogenic Shock at the time of index evaluation. The clinical and hemodynamic criteria used to diagnose Cardiogenic Shock will be those as defined in the Society for Cardiovascular Angiography and Interventions clinical expert consensus statement on the classification of cardiogenic shock.

SUMMARY:
This large real-world international prospective registry will provide a unique opportunity to comprehensively understand the contemporary management, clinical course and short as well as long-term outcomes of all Cardiogenic Shock (CS) patients cared for at four high volume dedicated shock care centers. As the first true North American multicenter CS collaborative with a uniform dedicated and comprehensive case report form, the high patient volumes and wide spectrum of clinical acuity seen at these institutions will provide valuable insight into the factors associated with adverse outcomes; and will serve as a blueprint for future clinical trial designs that may better inform clinical practice.

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is a hemodynamically complex and morbid syndrome characterized by frank circulatory collapse and end organ malperfusion stemming from severely impaired myocardial contractility. Despite advances in early reperfusion and regionalized systems of care, it remains the leading cause of in-hospital death following acute myocardial infarction (AMI) to this day, with mortality rates in excess of 40%. CS is also multifactorial with etiologies that extend beyond the reaches of acute coronary thrombosis, as more than 60% of cases may be due to acute decompensated heart failure (ADHF), a heterogenous conglomeration of disease states that remain poorly understood with equally dismal outcomes. In addition, while there has been a growing interest and significant uptake in the utilization of percutaneous mechanical circulatory support devices (pMCS) capable of providing greater procedural hemodynamics compared to the traditional intra-aortic balloon pump (IABP), they have yet to demonstrate a survival benefit.

In the absence of randomized trials to inform clinical care, there has been a growing interest in the development of an algorithmic approach to guide CS management, predicated on: 1) Early disease recognition; 2) Classification using a standardized nomenclature that incorporates comprehensive hemodynamics; 3) Selective and phenotypically tailored selective circulatory support; and 4) Multidisciplinary team-based care. While preliminary short-term results from United States CS registries employing such an approach has been favorable, there remain gaps in knowledge regarding a number of clinical domains in CS care, including: 1) Prognostic validation of invasive hemodynamics and risk stratification tools at the time of diagnosis; 2) Best practices for revascularization using contemporary therapies for AMI-CS patients; 3) Clinical predictors of outcomes among the different severity stages of CS; 4) Potential merits of varying care models (hub-and-spoke networks, high intensity cardiac intensive care units; 5) Ideal weaning strategies for peripheral mechanical circulatory support (pMCS) devices; and 6) Intermediate and long-term outcomes following the index clinical event, including health-related quality of life measures in this highly frail and vulnerable patient population.

This registry will prospectively and retrospectively follow all patients admitted to their respective health care systems with the primary diagnosis of CS. Unlike other registries, patients will be followed even if mechanical circulatory support is not implemented. Each patient will be followed from time of hospital admission to disposition, and at 30 days, 6 months and 1 year following discharge. A comprehensive and detailed evaluation of each patient and de-identified variables will be collected during these time periods, including baseline demographics, index and serial hemodynamic/metabolic assessments, and clinical care during the longitudinal hospital course. Data will be collected regarding revascularization strategies, vasopressor dosing and pMCS device utilization, to include weaning and escalation strategies. Information will also be collected regarding any morbidities sustained during the course of care, both in the cardiac intensive care unit (CICU) and during the post-ICU course. These include major bleeding, vascular complications requiring surgical or endovascular therapy, device-related hemolysis, need for renal replacement therapy and stroke. Among patients surviving the index hospitalization, they will also undergo cognitive and health-related quality of life evaluations using validated instruments at 30 days, 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of cardiogenic shock at time of index evaluation; including acute myocardial infarction- and acute decompensated heart failure-cardiogenic shock phenotypes
* Patients with cardiac arrest complicating cardiogenic shock and those with massive pulmonary embolism with right ventricular cardiogenic shock will also be eligible for the registry

Exclusion Criteria:

* Patients with shock not due to primary cardiac etiology will be excluded. These include septic, hemorrhagic, and anaphylactic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with cardiogenic shock at one of four high-volume North American quaternary care centers (Inova Heart and Vascular Institute, Sentara Norfolk General Hospital, University of Toronto and University of Utah)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  Percentage of participants alive at analysis time points

SECONDARY OUTCOMES:
Vascular Complications | 1 year
  Percentage of participants experiencing stroke or need for renal replacement therapy
Major Adverse Cardiovascular and Cerebrovascular Events | 1 year
  Percentage of participants experiencing myocardial infarction, stroke or heart failure re-hospitalization
Neurologic Status | 1 year
  Average participant neurologic status, as determined by the Cerebral Performance Category instrument
Health-related Quality of Life | 1 year
  Average participant health-related quality of life score, using the Rand 36-Item Short Form Survey

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Drakos, M.D., Principal Investigator — University of Utah
Locations (3):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Inova Heart and Vascular Institute, Falls Church, Virginia
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No